CLINICAL TRIAL: NCT04259099
Title: Validation of the Turkish Version of Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 (QUALEFFO-31)
Brief Title: Validation of the Turkish Version of QUALEFFO-31
Status: Terminated | Type: Observational
Why Stopped: Except in compulsory cases hospital admissions have been decreased significantly due to the pandemic. The study was terminated due to significant decrease in enrollment rate.
Sponsor: Bugra Ince (Other)
Responsible Party: Sponsor-Investigator, Bugra Ince, Medical Doctor, Principal Investigator, Bezmialem Vakif University
Organization: Bezmialem Vakif University (Other)
Other Study IDs: 54022451-050.05.04-01/16
Record Dates: First submitted 2020-02-02; First posted 2020-02-06 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Osteoporosis
Keywords: osteoporosis; Questionnaire; Quality of Life; QUALEFFO
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- QUALITY OF LIFE QUESTIONNAIRES: The group is anticipated to consist of 150 female and male with osteoporosis, osteopenia or normal bone mineral density.
  Interventions: Other: Testing the Quality of Life Questionnaire of the European Foundation for Osteoporosis-31(QUALEFFO-31)

INTERVENTIONS:
Other: Testing the Quality of Life Questionnaire of the European Foundation for Osteoporosis-31(QUALEFFO-31) — Administer the questionnaires to 150 participants to classify their status of quality of life.
  Other Names: Testing the Short Form-36 (SF-36)

SUMMARY:
The aim of this study is to investigate the adaptation and validity of the Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 in patients with osteoporosis. Thus, to present a scale that will help us analyze the psychometric properties of patients with osteoporosis to the use of the Turkish people .

DETAILED DESCRIPTION:
Osteoporosis has become an important public health problem due to low bone mass, decreased bone strength and increased risk of fractures. Today, the measurement of quality of life plays an important role in the approach to diseases. Quality of Life Questionnaire of the European Foundation for Osteoporosis-41 (QUALEFFO-41) has been used for many years as a well-established and fully self-administered questionnaire. In the following years, a shorter and more practical version was needed because the QUALEFFO-41 contains many questions and takes a long time. For this reason, the questionnaire was updated in 2006 and the version of QUALEFFO-31 was made and the validity of the current questionnaire was shown. The aim of this study is to conduct the reliability and validity study of Turkish version of QUALEFFO-31 and to evaluate the power of the questionnaire to distinguish patients with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* To have Dual-energy X-ray absorptiometry (DXA) results and thoracolumbar lateral spine X-Rays taken for any reason in the last 6 months.
* To have calcium, phosphorus, parathormone (PTH) and 25-hydroxyvitamin D level in the last 3 months.
* To be independently ambulatory.
* To have a cognitive capacity to understand and complete the questionnaires.

Exclusion Criteria:

* To have malignancy.
* To have inflammatory diseases.
* To have a metabolic bone disease other than osteoporosis.
* To have neuromuscular diseases.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females and males aged 50 and older with osteoporosis, osteopenia or normal bone mineral density.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Reliability and validity of the Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 | Through study completion, an average of 6 months
  Internal consistency will be tested with Cronbach Alpha coefficient. Intergroup reliability and consistency will be evaluated by T-Test.
Correlation between Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 and Short Form-36. | Through study completion, an average of 6 months
  The Spearman Correlation Analysis will be used for the correlation between QUALEFFO-31 and SF-36.
Testing Short Form-36 | Through study completion, an average of 6 months
  SF-36 is a self-assessment instrument. It consists of eight domains: bodily pain, physical functioning, social functioning, general health, mental health, vitality, and role restrictions due to physical and emotional problems.SF-36 is scored from 0 to 100. 0 indicated poor health status and 100 indicated good health status.
Testing Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 | Through study completion, an average of 6 months
  QUALEFFO-31 is a self-assessment instrument. It consists of three domains: pain,physical function and a mental function. QUALEFFO-31 is scored from 0 to 100. Domain scores were calculated by summing the scores of questions included in the domain and submitting the sum to a linear transformation to a scale of 100. Zero indicated good health status and 100 indicated poor health status.

CONTACTS AND LOCATIONS:
Overall Officials: Bugra Ince, MD, Principal Investigator — Bezmialem Vakif University Hospital
Locations (1):
- Bezmialem Vakif University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Schoor NM, Knol DL, Glas CA, Ostelo RW, Leplege A, Cooper C, Johnell O, Lips P. Development of the Qualeffo-31, an osteoporosis-specific quality-of-life questionnaire. Osteoporos Int. 2006;17(4):543-51. doi: 10.1007/s00198-005-0024-7. Epub 2005 Dec 14. PMID 16362146
- [Background] Lips P, Cooper C, Agnusdei D, Caulin F, Egger P, Johnell O, Kanis JA, Kellingray S, Leplege A, Liberman UA, McCloskey E, Minne H, Reeve J, Reginster JY, Scholz M, Todd C, de Vernejoul MC, Wiklund I. Quality of life in patients with vertebral fractures: validation of the Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO). Working Party for Quality of Life of the European Foundation for Osteoporosis. Osteoporos Int. 1999;10(2):150-60. doi: 10.1007/s001980050210. PMID 10501796
- [Derived] Ince B, Kucukakkas O. The reliability and validity of the Turkish version of the Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 (QUALEFFO-31). Arch Osteoporos. 2021 Sep 9;16(1):128. doi: 10.1007/s11657-021-00997-4. PMID 34499238